CLINICAL TRIAL: NCT06778954
Title: Prospective Randomized Controlled Trial of Ropivacaine-Poloxamer 407 Based Gel Application on Postoperative Pain After Open Gastrectomy
Brief Title: Ropivacaine-Poloxamer 407 Gel for Pain Control After Open Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2024-0383
Record Dates: First submitted 2025-01-05; First posted 2025-01-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peritoneal application group (Experimental): Patients who applied Ropivacaine-Poloxamer 407 hydrogel on space between peritoneum and fascia
  Interventions: Procedure: Arm I (Peritoneal application group)
- Subcutaneous injection group (Experimental): Patients who injected Ropivacaine-Poloxamer 407 hydrogel on subcutaneous area
  Interventions: Procedure: Arm II (Subcutaneous injection group)
- Placebo group (Placebo Comparator): Patients who did not apply Ropivacaine-Poloxamer 407 hydrogel
  Interventions: Procedure: Arm I (Peritoneal application group); Procedure: Arm II (Subcutaneous injection group)

INTERVENTIONS:
Procedure: Arm I (Peritoneal application group) — At the end of gastrectomy, during closure of incision, peritoneum and fascia are closed by suture, layer by layer. Skin approximation is doen with skin stapler. Ropivacaine-Poloxamer 407 hydrogel is applied on space between peritoneum and fascia in Arm I.
  Arms: Peritoneal application group; Placebo group
Procedure: Arm II (Subcutaneous injection group) — At the end of gastrectomy, during closure of incision, peritoneum and fascia are closed by suture, layer by layer. Skin approximation is doen with skin stapler. Ropivacaine-Poloxamer 407 hydrogel is injected on subcutaneous area in Arm II.
  Arms: Placebo group; Subcutaneous injection group

SUMMARY:
The study evaluates the efficacy of Ropivacaine-Poloxamer 407 hydrogel in reducing postoperative pain following open gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically confirmed diagnosis of gastric adenocarcinoma prior to surgery.
2. Patients who have undergone a complete surgical resection (R0 resection).
3. Patients with an ASA (American Society of Anesthesiologists) score of 3 or below.
4. Patients aged 20 years or older.

Exclusion Criteria:

1. Patients under 19 years of age.
2. Presence of ascites or peritoneal metastasis.
3. Patients who have undergone preoperative chemotherapy or radiotherapy.
4. Diagnosis of malignancies other than gastric cancer.
5. Uncontrolled diabetes, autoimmune diseases, hypertrophic scars, or keloid history affecting wound healing.
6. History of allergy or adverse reactions to Ropivacaine or other local anesthetics.
7. Pregnant women.
8. Patients with preoperative chronic pain conditions, including CRPS.
9. Patients with long-term preoperative use of opioid analgesics.
10. Patients with psychiatric disorders deemed likely to interfere with study participation.
11. Patients with severe liver disease, renal disease, or arrhythmia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total fentanyl consumption within 72 hours postoperatively. | Total fentanyl consumption within 72 hours postoperatively.
  The total amount of fentanyl administered to the patient via IV PCA during the initial 72-hour postoperative period will be recorded and compared among groups to assess analgesic efficacy.

SECONDARY OUTCOMES:
Pain intensity scores (NRS) at rest and during movement. | Pain intensity: Measured at 24, 48, and 72 hours postoperatively.
  Pain intensity: Numerical Rating Scale (NRS) scores ranging from 0 (no pain) to 10 (worst pain) assessed both at rest and during movement.
Time to first flatus and bowel movement. | Bowel function: Time to first flatus and bowel movement recorded until discahrge (within 6 days)
  Bowel function: Time to resume normal gastrointestinal activity.
Occurrence of postoperative nausea and vomiting (PONV). | PONV: Assessed daily for 72 hours.
  PONV: Incidence of nausea and vomiting documented along with severity scores.
Wound healing assessment, including seroma and infection rates. | Wound healing: Evaluated at regular intervals until first outpatient day (within 14 days)
  Wound healing: Observation of seroma or infection at the surgical site.
Length of hospital stay. | Hospital stay: up to 1 month
  Hospital stay: Measured in days from surgery until patient discharge.
Quality of recovery (QoR-15). | QoR-15: Measured at baseline and 72 hours postoperatively.
  QoR-15: Recovery quality assessed using a validated 15-item questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea